

1

## A Multicentre Observational Study to Evaluate Clinical Outcomes of the G7<sup>™</sup> Acetabular System

Protocol number: ORTHO.CR.GH20.13

Protocol date: 26 June 2013

NCT number: NCT02036931

G7 Early Evaluator



## 1 STUDY SYNOPSIS

| Complete Protocol Title | A Multicentre Observational Study to Evaluate Clinical Outcomes of the G7 <sup>™</sup> Acetabular System |
|---|---|
| Protocol Number | ORTHO.CR.GH20.13 |
| Short Protocol Title | G7 Early Evaluator |
| Sponsor | Zimmer GmbH |
| Manufacturer | Biomet Inc.; Biomet UK Ltd |
| Study Device(s) | G7 Acetabular Cup System |
| | The purpose of this multicenter study is to document the Clinical and Radiographic performance of the cup in both primary and revision procedures at the follow-up time points of 3 months, 1 year, 2 years, and 5 years and to report safety and Survivorship at 7 and 10 years follow-up. |
| | Primary endpoint: Harris Hip Score (HHS) at 2 year postoperative |
| Study Objectives/Endpoints | Secondary endpoints: |
| | a. Oxford Hip Score at 1,2,5 year postop |
| | b. Radiographic Evaluation: radiographic outcome, stability, incidence of radiolucencies around the prosthesis and bone remodeling |
| | c. Adverse Events/Complications (including revisions/removals of the study hip). d. Survivorship |
| Indications/Target Population | Subjects who have received G7 with one of three articulations (MOP, COP, COC) in primary or revision procedure and match with the indications for use. |
| Inclusion/Exclusion Criteria | <ul> <li>Inclusion Criteria</li> <li>Selection of subjects for this evaluation should be in accordance with the indications of the G7 cup specifically:</li> <li>Subjects with one of the following indication: <ul> <li>Noninflammatory degenerative joint disease including osteoarthritis and avascular necrosis.</li> <li>Rheumatoid arthritis.</li> <li>Correction of functional deformity.</li> <li>Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques.</li> <li>Revision procedures where other treatment or devices have failed.</li> </ul> </li> </ul> |



| | Additional inclusion criteria include: |
|---|---|
| | - Male or female. |
| | - 18 years of age or older |
| | - Subjects willing to return for follow-up evaluations. Subjects who read, understand study information and give written consent (specific local regulatory) |
| | Exclusion Criteria |
| | Exclusion criteria should be in accordance with Contraindications for the G7 cup. |
| | Absolute contraindications include: infection, sepsis and osteomyelitis, |
| | Additional contraindications include: |
| | - Subjects unable to cooperate with and complete the study |
| | <ul> <li>Dementia and inability to understand and follow instructions</li> <li>Neurological conditions affecting movement</li> </ul> |
| | - Pregnancy |
| Study Design | Prospective/Retrospective Observational Multi-Center<br>Non-Controlled post market surveillance study |
| Clinical Phase | Post-market |
| Sample Size | A sample size of 101 per group gives 80% power to detect a difference in means for each of the three comparisons. |
| Length of Study | 11 years (1-year enrolment, with a follow-up of 10 years) |
| Materials and Methods | Case report forms will be completed either in-office or hospital at Pre-op, Intra-Operative, Immediate Post-Operative, and the 3 Months, 1, 2, 5, 7 and 10-year intervals. |
| Data Collection | Paper/Electronic |
| Statistical Reporting | Statistical analysis will be conducted by Zimmer Biomet or its designee. Survivorship will be evaluated using Kaplan-Meier. |
| Scores/Performance Assessments | (modified) Harris Hip Score, Oxford Hip Score,<br>Radiographic Evaluations |
| Standards | <ul> <li>The PMCF is compliant with the below:</li> <li>ISO 14155: 2020 - Clinical investigation of medical devices for human subjects - Good clinical practice.</li> <li>The Declaration of Helsinki (DoH) - Ethical principles for medical research involving human subjects.</li> </ul> |



| Study Funding | Funding for this clinical study is made available by Zimmer Biomet to support clinical data collection, IRB/EC review fees and other expenses associated with the conduct and execution of this study protocol as outlined in the fully executed Clinical Trial Agreement. |
|---|---|
|---|---|